CLINICAL TRIAL: NCT03053063
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Selonsertib in Subjects With Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis (NASH)
Brief Title: Safety and Efficacy of Selonsertib in Adults With Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis (NASH)
Acronym: STELLAR-4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early due to lack of efficacy based on the results of the Week 48 analysis as prespecified in the clinical study protocol.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-384-1944; 2016-004148-13 (EudraCT Number)
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — selonsertib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEL 6 mg (Experimental): Randomized Phase: SEL 6 mg plus placebo to match SEL 18 mg for up to 240 weeks.
  Open-Label (OL) Phase: Participants who experienced a hepatic clinical event during the randomized phase prior to completing the Week 240 visit, will be offered the option to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks inclusive of the Randomized Phase.
  Interventions: Drug: SEL; Drug: Placebo to match SEL 18 mg
- SEL 18 mg (Experimental): Randomized Phase: SEL 18 mg plus placebo to match SEL 6 mg for up to 240 weeks.
  Open-Label Phase: Participants who experienced a hepatic clinical event during the randomized phase prior to completing the Week 240 visit, will be offered the option to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks inclusive of the Randomized Phase.
  Interventions: Drug: SEL; Drug: Placebo to match SEL 6 mg
- Placebo (Placebo Comparator): Randomized Phase: Placebo to match SEL 6 mg plus placebo to match SEL 18 mg for up to 240 weeks.
  Open-Label Phase: Participants who experienced a hepatic clinical event during the randomized phase prior to completing the Week 240 visit, will be offered the option to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks inclusive of the Randomized Phase.
  Interventions: Drug: Placebo to match SEL 6 mg; Drug: Placebo to match SEL 18 mg

INTERVENTIONS:
Drug: SEL — Tablets administered orally once daily
  Other Names: selonsertib; GS-4997
  Arms: SEL 18 mg; SEL 6 mg
Drug: Placebo to match SEL 6 mg — Tablets administered orally once daily
  Arms: Placebo; SEL 18 mg
Drug: Placebo to match SEL 18 mg — Tablets administered orally once daily
  Arms: Placebo; SEL 6 mg

SUMMARY:
The primary objective of this study is to evaluate whether selonsertib (SEL; GS-4997) can cause fibrosis regression and reduce associated complications in adults with cirrhosis due to NASH.

ELIGIBILITY:
Key Inclusion Criteria:

* Liver biopsy consistent with NASH and cirrhosis (F4 fibrosis) according to the NASH Clinical Research Network (CRN) classification, in the opinion of the central reader
* Has the following laboratory parameters at the screening visit, as determined by the central laboratory:

  * Alanine aminotransferase (ALT) ≤ 8 x upper limit of normal (ULN)
  * Creatinine Clearance (CLcr) ≥ 30 milliliter/minute (mL/min), as calculated by the Cockcroft-Gault equation
  * HbA1c ≤ 9.5% (or serum fructosamine ≤ 381 micromole (μmol) if HbA1c is unable to be resulted)
  * International normalised ratio (INR) ≤ 1.4, unless due to therapeutic anti-coagulation
  * Platelet count ≥ 100,000/μL

Key Exclusion Criteria:

* Prior history of decompensated liver disease including clinical ascites, hepatic encephalopathy (HE), or variceal bleeding
* Child-Pugh (CP) score > 7, as determined at screening, unless due to therapeutic anti-coagulation
* Model for End-stage Liver Disease (MELD) score > 12, as determined at screening, unless due to therapeutic anti-coagulation
* Other causes of liver disease including, but not limited to, alcoholic liver disease, hepatitis B, hepatitis C, autoimmune disorders, drug-induced hepatotoxicity, Wilson disease, iron overload, and alpha-1-antitrypsin deficiency, based on medical history and/or centralized review of liver histology.
* History of liver transplantation
* Current or history of hepatocellular carcinoma (HCC)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 883 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (283):
- United States (128):
  - Institute of Liver Health, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Baptist Medical Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Southern California Research Center, Coronado, California
  - Fresno Clinical Research Center, Fresno, California
  - Scripps Clinical Research Services, La Jolla, California
  - University of California, San Diego (Altman Clinical and Translational Research Center), La Jolla, California
  - Ruane Clinical Research Group, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affair Greater Los Angeles Healthcare System, West Los Angeles VA Medical Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Huntington Medical Research Institutes (HMRI) Liver Center, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Research and Education, Inc., San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center - Sutter Pacific Medical Foundation San Francisco Center for Liver Disease Dept. of Transplant, San Francisco, California
  - eStudySite, San Francisco, California
  - University of California, San Francisco-Liver Clinic, San Francisco, California
  - Island View Gastroenterology Associates- Ventura, Ventura, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Integrity Clinical Research, LLC, Doral, Florida
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - Clinical Research of Homestead, Homestead, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Florida Hospital Transplant Institute, Orlando, Florida
  - IMIC Inc, Palmetto, Florida
  - South Florida Center of Gastroenterology, PA, Wellington, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Piedmont Transplant Institute, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Northwestern Memorial Hospital; Clinical Research Unit, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem - Glenbrook ACC, Glenview, Illinois
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Iowa Digestive Disease Center, P.C., Clive, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - University of Louisville Clinical Trials Unit, Louisville, Kentucky
  - Delta Research Partners, Bastrop, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ocshner Medical Center, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC (STAR), Ridgeland, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Rutgers New Jersey Medical School- Doctors Office Center, Newark, New Jersey
  - AccumetRx Clinical Research, Albuquerque, New Mexico
  - University of Buffalo, Clinical and Translational Research Center, Buffalo, New York
  - Northwell Health - Sandra Atlas Bass Center for Liver Diseases, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai Beth Israel, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - NC TraCS Institute- CTRC, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas HealthCare System Center for Liver Disease, Charlotte, North Carolina
  - Duke University Medical Center - Duke South Clinics, Durham, North Carolina
  - Cumberland Research Associates LLC, Fayetteville, North Carolina
  - Piedmont HealthCare, d/b/a Carolinas Center for Liver Disease, Huntersville, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State University, The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC - Center for Liver Diseases at the Thomas E. Starlz Institute, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, University Hospital, Charleston, South Carolina
  - Greenville Health System Gastroenterology and Liver Center, Greenville, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Methodist University Hospital/University of Tennessee Health Science Center, Office of Clinical Research, Memphis, Tennessee
  - Quality Medical Research PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center - Digestive Disease Center, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Pinnacle Clinical Research, PLLC, Austin, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - Smith Clinic, Houston, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - DHAT Research Institute, Richardson, Texas
  - American Research Corporation, The Texas Liver Institute, San Antonio, Texas
  - Intermountain Liver Disease and Transplant Clinic, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc. d/b/a Bon Secours Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason, Seattle, Washington
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Australia (13):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St. George's Hospital, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Alfred Health, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - Medizinische Universitat Graz, Universitatsklinik fue Innere Medizin, Graz
  - Allgemeines Krankenhaus Wien, Vienna
- Belgium (5):
  - CUB Hopital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires UCL Saint-Luc, Brussels
  - Az Maria Middelares Ghent, Ghent
  - UZ Leuven, Leuven
- Canada (15):
  - University of Calgary Liver Unit (Heritage Medical Research Clinic), Calgary, Alberta
  - GI Research, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - LAIR Centre, Vancouver, British Columbia
  - Gordon and Leslie Diamond Health Care Centre, Vancouver General Hospital, UBC Division of Gastroenterology, Vancouver, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - University of Manitoba, Health Sciences Centre, John Buhler Research Centre, Winnipeg, Manitoba
  - South Shore Medical Arts, Bridgewater, Nova Scotia
  - William Osler Health System-Brampton Civic Hospital, Brampton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Toronto Center for Liver Diseases (TCLD), Toronto General Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Chronic Viral Illness Service/Royal Victoria Hospital/McGill University Health Centre (MUHC), Montreal, Quebec
- France (16):
  - CHU Amiens Picardie, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble- Hopital Michallon, Grenoble
  - Centre Hospitalier Regional Universitaire- Hopital Claude Huriez, Lille
  - CHU de Limoges- Hopital Dupuytren- Federation Hepatologie, Limoges
  - Hopital de la Croix Rousse, Lyon
  - Hôpital Saint Joseph, Marseille
  - CHU de Montpellier, Hopital St Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nice- Hopital l'Archet 2, Nice
  - Hopital Cochin, Paris
  - Groupe Hospitalier Universitaire La Pitie Salpetriere, Paris
  - Hopital Beaujon, Pessac
  - Centre Hospitalier Universitaire de Strasbourg- Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse- Hopital Purpan, Toulouse
- Germany (5):
  - Uniklinik RWTH Aachen, Medizinische Klinik III, Aachen
  - Universitatsklinikum Bonn (AoR), Bonn
  - Universitatsklinikum Frankfurt der Goethe-Universitat, Frankfurt am Main
  - Universitatsklinikum Leipzig AoR, Leipzig
  - Johannes Gutenberg-Universitat, Mainz
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
- India (10):
  - Department of Hepatology PGIMER Chandigarh, Chandigarh
  - Global Clinical Reseaech Services PVT LTD, Hyderabad
  - Institute of Post Graduate Medical Education and Research (IPGMER), Kolkata
  - Dayanand Medical College & Hospital, Ludhiana
  - Kasturba Medical College Hospital, Mangalore
  - Institute of Liver Diseases, HPB Surgery and Transplant Global Hospitals, Mumbai
  - Midas Multispecialty Hospital, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Delhi
  - Institute of Liver & Biliary Sciences, New Delhi
- Israel (7):
  - Emek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Japan (29):
  - Fukui-Ken Saiseikai Hospital, Fukui
  - Kyushu University Hospital, Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Kanazawa University Hospital, Kanazawa
  - Nara Medical University Hospital, Kashihara
  - Toranomon Hospital Kajigaya, Kawasaki
  - Kumamoto Shinto General Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Toranomon Hospital, Minato
  - Miyazaki Medical Center Hospital, Miyazaki
  - Aichi Medical University Hospital, Nagakute
  - Nara City Hospital, Nara
  - Kawasaki Medical School General Medical Center, Okayama
  - Okayama University Hospital, Okayama
  - Hirakata Kohsai Hospital, Osaka
  - National Hospital Organization Nagasaki Medical Center, Ōmura
  - Saga University Hospital, Saga
  - Hokkaido University Hospital, Sapporo
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Tokyo Womens Medical University Hospital, Shinjuku
  - Saiseikai Suita Hospital, Suita
  - Osaka University Hospital, Suita
  - Ehime University Hospital, Tōno
  - Mie University Hospital, Tsu
  - Yamagata University Hospital, Yamagata
  - Yokohama City University Hospital, Yokohama
- Mexico (2):
  - Consultorio Médico, Mexico City
  - Accelerium S. de R.L. de C.V., Monterrey
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Southern District Health Board - Dunedin Hospital, Dunedin
- Poland (3):
  - Szpital Specjalistyczny Nr 1 w Bytomiu, Oddzial Obserwacyjno-Zakazny i Hepatologii, Bytom
  - Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego, Lodz
  - ID Clinic Arkadiusz Pisula, Mysłowice
- Puerto Rico (3):
  - Klinical Investigations Group, LLC, San Juan
  - VA Carribean Healthcare System, San Juan
  - Fundacion de Investigacion de Diego, San Juan
- Singapore (3):
  - National University Health System, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital Pte Ltd., Singapore
- South Korea (10):
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - National Health Insurance Service- Ilsan Hospital, Goyang-si
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (11):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar - Parc de Salut, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerto de Hierro Majadahonda, Majadahonda
  - CHOP_Complejo Hospitalario Universitario de Pntevedra, Pontevedra
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Switzerland (2):
  - Universitätsklinik für Viszerale Chirurgie und Medizin, Inselspital, Hepatologie, Bern
  - Istituto Cantanale di Patologia Locarno, Lugano
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-LinKou Branch, Taoyuan District
- United Kingdom (9):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Barts Health NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St. George's Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Plymouth Hospitals NHS Trust, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Abertawe Bro Morgannwg University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Anstee QM, Lawitz EJ, Alkhouri N, Wong VW, Romero-Gomez M, Okanoue T, Trauner M, Kersey K, Li G, Han L, Jia C, Wang L, Chen G, Subramanian GM, Myers RP, Djedjos CS, Kohli A, Bzowej N, Younes Z, Sarin S, Shiffman ML, Harrison SA, Afdhal NH, Goodman Z, Younossi ZM. Noninvasive Tests Accurately Identify Advanced Fibrosis due to NASH: Baseline Data From the STELLAR Trials. Hepatology. 2019 Nov;70(5):1521-1530. doi: 10.1002/hep.30842. Epub 2019 Aug 19. PMID 31271665
- [Result] Alkhouri N, Younossi ZM, Lawitz EJ, Wong VWS, Romero-Gomez M, et al. Impact of age on routinely available noninvasive tests for the discrimination of advanced fibrosis due to NASH in the phase 3 STELLAR trials of the ASK1 inhibitor selonsertib [Poster SAT-273]. European Association for the Study of the Liver (EASL); 2019; Vienna Austria.
- [Result] Younossi ZM, Stepanova M, Anstee QM, Lawitz EJ, Wai-Sun Wong V, Romero-Gomez M, Kersey K, Li G, Subramanian GM, Myers RP, Djedjos CS, Okanoue T, Trauner M, Goodman Z, Harrison SA. Reduced Patient-Reported Outcome Scores Associate With Level of Fibrosis in Patients With Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2019 Nov;17(12):2552-2560.e10. doi: 10.1016/j.cgh.2019.02.024. Epub 2019 Feb 16. PMID 30779990
- [Result] Anstee QM, Lawitz EJ, Alkhouri N, Wai Sun Wong V, Romero-Gomez M, et al. Routinely available noninvasive tests discriminate advanced fibrosis due to NASH in the Phase 3 STELLAR trials of the ASK1 inhibitor selonsertib [poster]. American Association for the Study of Liver Diseases (AASLD); 2018, San Francisco, CA.
- [Result] Younossi ZM, Lawitz E, Alkhouri N, Wong VWS, Romero-Gomez M, et al. Algorithms using noninvasive tests can accurately identify patients with advanced fibrosis due to NASH: Data From the STELLAR clinical trials [Poster LB-10]. AASLD; 2018; San Francisco, CA.
- [Result] Younossi ZM, Stepanova M, Anstee QM, Lawitz EJ, Wai-Sun Wong V, et al. Severe impairment of patient-reported outcomes in patients with advanced fibrosis due to non-alcoholic steatohepatitis (NASH) [Poster]. AASLD; 2018; San Francisco, CA.
- [Result] Younossi ZM, Stepanova M, Anstee QM, Lawitz EJ, Wai Sun Wong V, et al. Advanced fibrosis based on noninvasive tests in nonalcoholic steatohepatitis (NASH) is associated with impairment of patient-reported outcomes [Poster]. AASLD; 2018; San Francisco, CA.
- [Result] Harrison SA, Wong VW, Okanoue T, Bzowej N, Vuppalanchi R, Younes Z, Kohli A, Sarin S, Caldwell SH, Alkhouri N, Shiffman ML, Camargo M, Li G, Kersey K, Jia C, Zhu Y, Djedjos CS, Subramanian GM, Myers RP, Gunn N, Sheikh A, Anstee QM, Romero-Gomez M, Trauner M, Goodman Z, Lawitz EJ, Younossi Z; STELLAR-3; STELLAR-4 Investigators. Selonsertib for patients with bridging fibrosis or compensated cirrhosis due to NASH: Results from randomized phase III STELLAR trials. J Hepatol. 2020 Jul;73(1):26-39. doi: 10.1016/j.jhep.2020.02.027. Epub 2020 Mar 6. PMID 32147362
- [Derived] Loomba R, Huang DQ, Sanyal AJ, Anstee QM, Trauner M, Lawitz EJ, Ding D, Ma L, Jia C, Billin A, Huss RS, Chung C, Goodman Z, Wong VW, Okanoue T, Romero-Gomez M, Abdelmalek MF, Muir A, Afdhal N, Bosch J, Harrison S, Younossi ZM, Myers RP. Liver stiffness thresholds to predict disease progression and clinical outcomes in bridging fibrosis and cirrhosis. Gut. 2023 Mar;72(3):581-589. doi: 10.1136/gutjnl-2022-327777. Epub 2022 Sep 9. PMID 36750244
- [Derived] Younossi ZM, Anstee QM, Wai-Sun Wong V, Trauner M, Lawitz EJ, Harrison SA, Camargo M, Kersey K, Subramanian GM, Myers RP, Stepanova M. The Association of Histologic and Noninvasive Tests With Adverse Clinical and Patient-Reported Outcomes in Patients With Advanced Fibrosis Due to Nonalcoholic Steatohepatitis. Gastroenterology. 2021 Apr;160(5):1608-1619.e13. doi: 10.1053/j.gastro.2020.12.003. Epub 2020 Dec 8. PMID 33307033
- [Derived] Younossi ZM, Stepanova M, Younossi I, Racila A. Validation of Chronic Liver Disease Questionnaire for Nonalcoholic Steatohepatitis in Patients With Biopsy-Proven Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2093-2100.e3. doi: 10.1016/j.cgh.2019.01.001. Epub 2019 Jan 11. PMID 30639779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Asia, Australia, New Zealand, Europe and Puerto Rico. The first participant was screened on 30 January 2017. The last study visit occurred on 06 May 2019.
Pre-assignment Details: 2154 participants were screened.
Groups:
- SEL 18 mg: Randomized Phase: Selonsertib (SEL) 18 mg tablet orally once daily + placebo for up to 240 weeks.
- SEL 6 mg: Randomized Phase: SEL 6 mg tablet orally once daily + placebo for up to 240 weeks.
- Placebo: Randomized Phase: Placebo to match SEL 18 mg and 6 mg tablets orally once daily for up to 240 weeks.
- Open-Label SEL 18 mg: Open-label (OL) Phase: Participants who experienced a hepatic clinical event during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration of 240 weeks, including the treatment duration in the randomized phase.
Period: Randomized Phase
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Open-Label SEL 18 mg
Started | 355 | 354 | 174 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 355 | 354 | 174 | 0
Not completed — Study Terminated by Sponsor | 326 | 317 | 161 | 0
Not completed — Withdrew consent | 8 | 11 | 5 | 0
Not completed — Investigator's Discretion | 8 | 6 | 2 | 0
Not completed — Lost to Follow-up | 3 | 5 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Randomized but Never Treated | 1 | 3 | 2 | 0
Not completed — Entered the Open-Label Phase | 9 | 11 | 3 | 0
Period: Open-Label Phase
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Open-Label SEL 18 mg
Started | 0 | 0 | 0 | 23 (Participants who experienced a hepatic clinical event had the option to roll over into the OL Phase.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 23
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 19
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Investigator's discretion | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- SEL 18 mg: Randomized Phase: SEL 18 mg tablet orally once daily + placebo for up to 240 weeks.
  Open-label Phase: Participants who experienced a hepatic clinical event during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration, including the treatment duration in the randomized phase, of 240 weeks.
- SEL 6 mg: Randomized Phase : Selonsertib (SEL) 6 mg tablet orally once daily + placebo for up to 240 weeks.
  Open-label (OL) Phase: Participants who experienced a hepatic clinical event during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an open-label phase to receive OL SEL 18 mg daily for a total treatment duration, including the treatment duration in the randomized phase, of 240 weeks.
- Placebo: Randomized Phase: Placebo tablet orally once daily for up to 240 weeks.
  Open-label Phase: Participants who experienced a hepatic clinical event during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration, including the treatment duration in the randomized phase, of 240 weeks.
- Total: Total of all reporting groups
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Total
Number analyzed (Participants) | 354 | 351 | 172 | 877
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8.5) | 57 (8.7) | 60 (8.4) | 58 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 230 | 101 | 547
  Male | 138 | 121 | 71 | 330
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 3 | 3 | 0 | 6
  Race: Asian | 73 | 59 | 33 | 165
  Race: Black | 5 | 4 | 1 | 10
  Race: Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 1
  Race: White | 261 | 279 | 136 | 676
  Race: Other | 7 | 6 | 1 | 14
  Race: Not Permitted | 4 | 0 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 300 | 297 | 149 | 746
  Ethnicity: Hispanic or Latino | 49 | 51 | 22 | 122
  Ethnicity: Not Permitted | 5 | 3 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a ≥ 1-Stage Improvement in Fibrosis According to the Nonalcoholic Steatohepatitis (NASH) Clinical Research Network (CRN) Classification Without Worsening of NASH
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH CRN classification. NASH CRN fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis). Worsening of NASH was defined as ≥ 1 point increase from baseline in hepatocellular ballooning or lobular inflammation according to the Non-Alcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) criteria. As defined by NAS, hepatocellular ballooning ranges from 0-2 and lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation.
Time Frame: Week 48
Population: The Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 354 | 351 | 172
percentage of participants | 14.4 [10.9 to 18.5] | 12.8 [9.5 to 16.8] | 12.8 [8.2 to 18.7]
Statistical Analysis 1: Comparison: SEL 18 mg vs Placebo; Test type: Superiority; p = 0.5572, Mantel Haenszel — Difference between SEL 18 mg vs Placebo, 95% confidence interval (CI) and p-value were obtained by stratified Mantel-Haenszel method adjusting for baseline (BL) diabetes mellitus status and BL Enhanced Liver Fibrosis (ELF) score (<11.27 vs ≥11.27); Percentage Difference = 1.9, 95% CI 2-sided [-4.4 to 8.2]
Statistical Analysis 2: Comparison: SEL 6 mg vs Placebo; Test type: Superiority; p = 0.9272, Mantel Haenszel — Difference between SEL 6 mg vs Placebo, 95% CI and p-value were obtained by stratified Mantel-Haenszel method adjusting for BL diabetes mellitus status and BL ELF score (<11.27 vs ≥11.27); Percentage Difference = 0.3, 95% CI 2-sided [-6.0 to 6.5]

2. Primary Outcome: Event-Free Survival (EFS) at Week 240 as Assessed by Time to First Clinical Event
Description: EFS was assessed by the time to the first clinical event, including liver decompensation events, liver transplantation and all-cause mortality.
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Had a ≥ 1-Stage Improvement in Fibrosis Without Worsening of NASH at Week 240
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH CRN classification. NASH CRN fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis). Worsening of NASH was defined as ≥ 1 point increase from baseline in hepatocellular ballooning or lobular inflammation according to the NAS criteria. As defined by NAS, hepatocellular ballooning ranges from 0-2 and lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation.
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Who Had a ≥ 1-Stage Improvement in Fibrosis at Week 48
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH CRN classification. NASH CRN fibrosis stages range from 0 to 4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis).
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 354 | 351 | 172
percentage of participants | 18.9 [15.0 to 23.4] | 16.8 [13.0 to 21.1] | 15.7 [10.6 to 22.0]
Statistical Analysis 1: Comparison: SEL 18 mg vs Placebo; Test type: Superiority; p = 0.2850, Mantel Haenszel — Difference between SEL 18 mg vs Placebo, 95% CI and p-value were obtained by stratified Mantel-Haenszel method adjusting for BL diabetes mellitus status and BL ELF score (<11.27 vs ≥11.27); Percentage Difference = 3.8, 95% CI 2-sided [-3.1 to 10.6]
Statistical Analysis 2: Comparison: SEL 6 mg vs Placebo; Test type: Superiority; p = 0.6731, Mantel Haenszel — [p-value comment as in outcome 1, analysis 2]; Percentage Difference = 1.5, 95% CI 2-sided [-5.3 to 8.2]

5. Secondary Outcome: Percentage of Participants Who Had a ≥ 1-Stage Improvement in Fibrosis at Week 240
Description: as for outcome 4
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Had NASH Resolution at Week 48
Description: NASH resolution was defined as lobular inflammation of 0 or 1 from ≥ 1 at baseline and hepatocellular ballooning reduced to 0 from a value ≥ 1 at baseline; both criteria were necessary conditions. As defined by NAS, hepatocellular ballooning ranges from 0-2 and lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation. Evaluable participants had baseline lobular inflammation and hepatocellular ballooning ≥ 1.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 353 | 351 | 172
percentage of participants | 2.3 [1.0 to 4.4] | 3.7 [2.0 to 6.3] | 4.1 [1.7 to 8.2]
Statistical Analysis 1: Comparison: SEL 18 mg vs Placebo; Test type: Superiority; p = 0.3650, Mantel Haenszel — [p-value comment as in outcome 4, analysis 1]; Percentage Difference = -1.7, 95% CI 2-sided [-5.5 to 2.0]
Statistical Analysis 2: Comparison: SEL 6 mg vs Placebo; Test type: Superiority; p = 0.8557, Mantel Haenszel — [p-value comment as in outcome 1, analysis 2]; Percentage Difference = -0.4, 95% CI 2-sided [-4.3 to 3.6]

7. Secondary Outcome: Percentage of Participants Who Had NASH Resolution at Week 240
Description: NASH resolution was defined as lobular inflammation of 0 or 1 from ≥ 1 at baseline and hepatocellular ballooning reduced to 0 from a value ≥ 1 at baseline; both criteria were necessary conditions.As defined by NAS, hepatocellular ballooning ranges from 0-2 and lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation. Evaluable participants had baseline lobular inflammation and hepatocellular ballooning ≥ 1.
Time Frame: Week 240
Population: No data was analyzed as the study was terminated and no participants reached the Week 240 timepoint.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose date up to last dose (maximum: 108.7 weeks) plus 30 days
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- SEL 18 mg: Randomized Phase: SEL 18 mg tablet orally once daily + placebo for up to 240 weeks.
- Placebo: Randomized Phase: Placebo tablet orally once daily for up to 240 weeks.
- Open-Label SEL 18 mg: Participants who experienced a hepatic clinical event during the randomized phase, prior to completing the Week 240 visit, were offered the option to roll over into an OL phase to receive OL SEL 18 mg daily for a total treatment duration, including the treatment duration in the randomized phase, of 240 weeks.
Arm/Group | SEL 18 mg | SEL 6 mg | Placebo | Open-Label SEL 18 mg
All-Cause Mortality (participants affected / at risk) | 0/354 | 0/351 | 0/172 | 2/23
Serious Adverse Events (participants affected / at risk) | 60/354 | 53/351 | 22/172 | 7/23
Other Adverse Events (participants affected / at risk) | 251/354 | 276/351 | 135/172 | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEL 18 mg (N=354) | SEL 6 mg (N=351) | Placebo (N=172) | Open-Label SEL 18 mg (N=23)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Visceral venous thrombosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 3 | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 2 | 3 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 3 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Haemobilia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Intrahepatic portal hepatic venous fistula (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 3 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Model for end stage liver disease score increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 2 | 1 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometrial thickening (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hydrosalpinx (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEL 18 mg (N=354) | SEL 6 mg (N=351) | Placebo (N=172) | Open-Label SEL 18 mg (N=23)
Abdominal distension (Gastrointestinal disorders) | 22 | 22 | 12 | 3
Abdominal pain (Gastrointestinal disorders) | 34 | 33 | 19 | 2
Abdominal pain upper (Gastrointestinal disorders) | 42 | 37 | 21 | 3
Constipation (Gastrointestinal disorders) | 46 | 47 | 18 | 0
Diarrhoea (Gastrointestinal disorders) | 51 | 60 | 40 | 2
Nausea (Gastrointestinal disorders) | 47 | 59 | 17 | 2
Vomiting (Gastrointestinal disorders) | 24 | 28 | 7 | 3
Fatigue (General disorders) | 42 | 51 | 20 | 0
Oedema peripheral (General disorders) | 20 | 23 | 10 | 1
Bronchitis (Infections and infestations) | 16 | 27 | 10 | 0
Influenza (Infections and infestations) | 27 | 24 | 8 | 1
Nasopharyngitis (Infections and infestations) | 42 | 33 | 28 | 0
Sinusitis (Infections and infestations) | 25 | 27 | 11 | 1
Upper respiratory tract infection (Infections and infestations) | 43 | 52 | 15 | 1
Urinary tract infection (Infections and infestations) | 33 | 39 | 11 | 0
Procedural pain (Injury, poisoning and procedural complications) | 20 | 23 | 12 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 28 | 15 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 30 | 16 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 25 | 10 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 19 | 9 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 19 | 5 | 1
Dizziness (Nervous system disorders) | 22 | 23 | 17 | 1
Headache (Nervous system disorders) | 47 | 48 | 21 | 4
Hepatic encephalopathy (Nervous system disorders) | 7 | 5 | 2 | 4
Insomnia (Psychiatric disorders) | 24 | 28 | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 33 | 14 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 27 | 11 | 2
Rash (Skin and subcutaneous tissue disorders) | 19 | 13 | 10 | 1

LIMITATIONS AND CAVEATS:
Based on the results of the Week 48 analysis, the study was terminated early for lack of efficacy as prespecified in the clinical study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03053063/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03053063/SAP_001.pdf